CLINICAL TRIAL: NCT01073137
Title: Noninvasive Blood Glucose Monitoring Using Otoacoustic Emissions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Eric A. Wan, Oregon Health & Sciences University
Other Study IDs: 1R21DK079283-01A1 (NIH)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic Subjects
- Non diabetic subjects

SUMMARY:
The purpose of the research is to determine whether a noninvasive hearing test may be used to predict blood glucose in people with diabetes.

DETAILED DESCRIPTION:
Participation in the study will involve listening to sounds through earphones while blood glucose levels are measured by taking blood samples using a lancet. During the study, blood glucose levels will be increased by drinking a beverage containing sugar.

Up to five visits to the NCRAR will be needed over a six-month period to complete the study. Each visit lasts either two or four hours, and will be scheduled at your convenience. You will be paid $20 for the first 2-hour screening visit and $50 for each 4-hour visit. You will be paid $30 if you are selected to participate in a 2-hour Attention Correlation Test that a sub-set of 10 participants will complete.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diabetes
* Normal hearing
* Hemoglobin A1C of 5.5-8%

Exclusion Criteria:

* Volunteers may not participate if they have peripheral neuropathy

  * visual impairment due to diabetic retinopathy
  * organ failure (kidney, liver heart, or lungs)
  * severe or unstable cardiovascular disease
  * active alcohol or drug abuse
  * schizophrenia
  * bipolar disorder
  * active major depressive disorder
  * active foot ulcerations
  * active viral or other infections such as HIV
  * hepatitis, or pneumonia
  * serious renal
  * cardiac or cognitive dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetese subjects with no hearing impairement.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Otoacoustic emissions change with blood sugar levels | One 2-hour screening visit, and on 4-hour visit

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Wan, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States